CLINICAL TRIAL: NCT01283230
Title: Prospective Cohort Study for Evaluation of Liver Fibrosis Staging With Acoustic Radiation Force Impulse Elastography in Patients With Chronic Liver Disease and Healthy Liver/Kidney Donors
Brief Title: Evaluation of Liver Fibrosis Staging With Acoustic Radiation Force Impulse Elastography
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2010-0015
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Liver Disease
Keywords: ARFI imaging; normal values; chronic liver disease; liver donors; kidney donors
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- chronic liver disease: Any cause of liver disease that involves a process of progressive destruction and regeneration of the liver parenchyma leading to fibrosis and cirrhosis such as hepatitis B, hepatitis C, alcoholic liver disease.
  Interventions: Device: Acoustic radiation force impulse imaging
- Healthy liver and kidney donor: Healthy liver and kidney donor who have normal liver condition
  Interventions: Device: Acoustic radiation force impulse imaging

INTERVENTIONS:
Device: Acoustic radiation force impulse imaging — Acoustic radiation force impulse (ARFI) imaging were measured 10 times in each patient.The region of interest was chosen in an area where the normal liver parenchyma was at least 6 cm thick and free of large blood vessels was chosen. A measurement depth of 2 cm below the liver capsule was chosen to standardize the examination.
  Other Names: ARFI imaging

SUMMARY:
This is a prospective cohort Study for evaluation of liver fibrosis staging with acoustic radiation force impulse elastography in patients with chronic liver disease and healthy liver/kidney donors.

DETAILED DESCRIPTION:
A recent new method for liver fibrosis assessment based on similar technology to transient elastography is acoustic radiation force impulse (ARFI) imaging. ARFI has the advantages which can be conducted in parallel ways of measuring points in the patients with chronic liver disease when they underwent routine ultrasound examination. Thus, the aim of this study was to identify the normal range of ARFI velocity and assess the best cut-off value by recruiting healthy living liver and kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* chronic liver disease (hepatitis B, hepatitis C, liver cirrhosis) patients who are planned to liver biopsy
* Healthy liver and kidney donors
* The patients who is willing and able to provide written informed consent to participate in this study

Exclusion Criteria:

* Decompensated liver cirrhosis
* Patients with liver congestion due to heart dysfunction
* Patients who previously take antiviral agent and antifibrotic agent
* Healthy liver and kidney donors with any laboratory abnormalities regarding liver condition (Platelet count < 150 x 103/ul, Fasting glucose > 110 mg/dl, AST > 40 IU/L, ALT> 40 IU/L, Albumin < 3.3 g/dl, Total bilirubin > 1.2 mg/dl, GGT> 54 IU/L, ALP > 115 IU/L , Ferritin > 322 ng/ml)
* A history of any other medical disease or condition that would make the patients unsuitable for this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease, Healthy liver and kidney donors
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of ARFI velocity in healthy donors and patients with chronic liver disease | 2 years
  Measurement of ARFI velocity is non-invsive ultrasonographic technique. It is performed with a abdominal convex probe which is same probe as conventional ultrasonography. Short-duration acoustic radiation forces result in shear-wave propagation away from the region of excitation and are tracked using ultrasonic correlation-based methods. This results are called ARFI velocity which is expressed as meters per second

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Hyub Han, MD, Study Chair — Department of Internal Medicine, Yonsei University College of Medicine; Seung Up Kim, MD, Principal Investigator — Department of Internal Medicine, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea